CLINICAL TRIAL: NCT01177904
Title: Early Progesterone Cessation After in Vitro Fertilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Graciela Kohls, Gynecologist, IVI Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAD-GK-01-2009-02
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Pregnant Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone 5 Weeks (Active Comparator): The study group stop receiving P4 on the day of their first US at 5 weeks pregnancy
  Interventions: Other: Cease progsterone at 5
- Control Group : P4 8 weeks (Other): Progesterone will be given until 8 weeks of pregnancy
  Interventions: Other: control group: progesterone 8

INTERVENTIONS:
Other: Cease progsterone at 5 — Cease administration of progsterone at first US at 5 weeks
  Arms: Progesterone 5 Weeks
Other: control group: progesterone 8 — Control group: progesterone until 8 weeks of pregnancy
  Arms: Control Group : P4 8 weeks

SUMMARY:
There seems to be a general consensus on the supplementation of progesterone (P4) for luteal phase support (LPS) to all women after in vitro fertilization (IVF) treatment. However, there is no agreement about the precise duration of LPS.

DETAILED DESCRIPTION:
The objective of the study is to investigate the effect of early cessation of progesterone for LPS after IVF treatment on the pregnancy outcome, with special interest in determining the miscarriage rate and episodes of bleeding between the date of the first ultrasound (US) and up to 12 weeks of gestation.

Patients start to receive 200 mg twice a day of P4 on the day after oocyte retrieval.

All patients which show a gestational sac in their uterus in the first US are included in this study and randomized.

Inclusion criteria:

1. Patients who underwent ovarian stimulation using GnRH analogues,
2. Fresh embryo transfer,
3. LPS by vaginal micronized P4,
4. Clinical pregnancy demonstrated by US and
5. Informed consent signed.

Exclusion criteria:

Patients who had bleeding episodes before their first US because they are likely to continue P4 therapy without medical indication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent ovarian stimulation using GnRH analogues,
2. Fresh embryo transfer,
3. LPS by vaginal micronized P4,
4. Clinical pregnancy demonstrated by US and
5. Informed consent signed.

Exclusion Criteria:

Patients who had bleeding episodes before their first US because they are likely to continue P4 therapy without medical indication.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Garcia-Velasco, MD, PhD, Study Director — IVI Madrid
Locations (1):
- IVI-Madrid, Madrid, Spain

REFERENCES:
- [Derived] Kohls G, Ruiz F, Martinez M, Hauzman E, de la Fuente G, Pellicer A, Garcia-Velasco JA. Early progesterone cessation after in vitro fertilization/intracytoplasmic sperm injection: a randomized, controlled trial. Fertil Steril. 2012 Oct;98(4):858-62. doi: 10.1016/j.fertnstert.2012.05.046. Epub 2012 Jun 29. PMID 22749223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Progesterone during 1st trimester
Groups:
- Progesterone 5 Weeks: The study group stop receiving progesterone on the day of their first Ultra-sound at 5 weeks pregnancy
  Cease progesterone at 5: Cease administration of progesterone at first Ultra-sound at 5 weeks
- Control Group : Progesterone 8 Weeks: Progesterone will be given until 8 weeks of pregnancy
  control group: progesterone 8: Control group: progesterone until 8 weeks of pregnancy
Period: Overall Study
Arm/Group | Progesterone 5 Weeks | Control Group : Progesterone 8 Weeks
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Women
Groups:
- Progesterone 5 Weeks: The study group of women stop receiving P4 on the day of their first US at 5 weeks pregnancy
  Cease progsterone at 5: Cease administration of progsterone at first US at 5 weeks
- Total: Total of all reporting groups
Arm/Group | Progesterone 5 Weeks | Control Group : P4 8 Weeks | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 200
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Bleeding Episodes [Mean (Standard Deviation); unit: Bleeding episodes] — Bleeding Episodes in each group.
  Bleeding episodes | 8 (4) | 8 (4) | 8 (4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeding Episodes
Description: Number of bleeding episodes up to a year
Time Frame: Up to year
Measure: Mean (Standard Deviation); unit: Episodes of bleeding
Groups:
- Study Group: The study group stop receiving progesterone on the day of their first Ultra-sound at 5 weeks pregnancy
  Cease progesterone at 5: Cease administration of progesterone at first Ultra-sound at 5 weeks
Arm/Group | Control Group : P4 8 Weeks | Study Group
Number analyzed (Participants) | 100 | 100
Episodes of bleeding | 8 (10) | 8 (10)

ADVERSE EVENTS:
Groups:
- Study Group: P4 5 Weeks: Progesterone will be given until 5 weeks of pregnancy
Arm/Group | Control Group : P4 8 Weeks | Study Group: P4 5 Weeks
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes